CLINICAL TRIAL: NCT00445289
Title: Automatic Control of Pressure Support Ventilation in Surgical Intensive Care Units - a Bicentric, Prospective, Randomized, Controlled Trial
Brief Title: Automatic Control of Pressure Support Ventilation in Surgical Intensive Care Units
Acronym: ASOPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASOPI
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2008-08-18 (Estimated); Status verified 2008-08

CONDITIONS: Ventilator Weaning
Keywords: mechanical ventilation; ventilator weaning; closed-loop; ventilation time

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: SmartCare/PS

SUMMARY:
This bicentric, randomized, controlled trial examines the effectiveness of an automatic control of pressure support ventilation (SmartCare/PS) in critically ill patients.

DETAILED DESCRIPTION:
During the weaning process vigilance, pulmonary mechanics and respiratory drive of the patient are changing. Consequently, ventilation settings have to be modified very often. The modifications can be conducted either according to a weaning protocol or automatically by an expert system (SmartCare/PS). This trial compares protocol-guided weaning with automatic weaning in post-surgical patients and examines the effect on total ventilation time, numbers of manipulations and alarms of the ventilator, length of stay in the ICU and in the hospital, 28- and 90-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* Intubated or tracheotomised patients requiring mechanical ventilation at 9:00 am for longer than 9 hours (within this time period invasive and non-invasive ventilation is permitted)

Exclusion Criteria:

* Cerebral trauma / surgery
* Age < 18 years
* Do-not-resuscitate-order
* Duration of mechanical ventilation > 24 h
* Patient is currently participating in this trial (including 90 days follow-up period)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Total ventilation time during intensive care unit stay.

SECONDARY OUTCOMES:
Time in the zone of respiratory comfort during invasive mechanical ventilation
Number of ventilator alarms during invasive mechanical ventilation
Number of ventilator manipulations during invasive mechanical ventilation
Length of ICU and hospital stay
28-day and 90-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jens Scholz, M.D., Principal Investigator — University Medical Centre Schleswig-Holstein, Campus Kiel, Department of Anaesthesiology and Intensive Care Medicine
Locations (2):
- Germany (2):
  - Department of Anaesthesiology and Intensive Care Medicine, Kiel
  - Department of Cardiovascular Surgery, Kiel

REFERENCES:
- [Background] Lellouche F, Mancebo J, Jolliet P, Roeseler J, Schortgen F, Dojat M, Cabello B, Bouadma L, Rodriguez P, Maggiore S, Reynaert M, Mersmann S, Brochard L. A multicenter randomized trial of computer-driven protocolized weaning from mechanical ventilation. Am J Respir Crit Care Med. 2006 Oct 15;174(8):894-900. doi: 10.1164/rccm.200511-1780OC. Epub 2006 Jul 13. PMID 16840741
- [Background] Dojat M, Brochard L, Lemaire F, Harf A. A knowledge-based system for assisted ventilation of patients in intensive care units. Int J Clin Monit Comput. 1992 Dec;9(4):239-50. doi: 10.1007/BF01133619. PMID 1484275
- [Derived] Schadler D, Engel C, Elke G, Pulletz S, Haake N, Frerichs I, Zick G, Scholz J, Weiler N. Automatic control of pressure support for ventilator weaning in surgical intensive care patients. Am J Respir Crit Care Med. 2012 Mar 15;185(6):637-44. doi: 10.1164/rccm.201106-1127OC. Epub 2012 Jan 20. PMID 22268137